CLINICAL TRIAL: NCT05572268
Title: IN VIVO AND IN VITRO COMPARATIVE STUDY ON EFFICACY OF ANSA (Experimental Drug) & CRAN MAX (Control Drug) SACHET IN UNCOMPLICATED UTI
Brief Title: EFFICACY OF ANSA (Experimental Drug) & CRAN MAX (Control Drug) SACHET
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shifa Ul Mulk Memorial Hospital (Other)
Responsible Party: Principal Investigator, Dr. Hafiz Muhammad Asif, Chairperson Department of Eastern Medicine, Jinnah University, Shifa Ul Mulk Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Misbah Ahmed; UTI (Other: Jinnah University)
Record Dates: First submitted 2022-09-28; First posted 2022-10-07 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Treatment Compliance
Keywords: Vaccinium macrocarpon, Saraca indica, Cimicifuga racemosa
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ANSA Sachet (Experimental): Ansa sachet having three APIs (Vaccinium macrocarpon, Saraca indica, Cimicifuga racemosa)
  Interventions: Drug: to evaluate the safety and efficacy of Ansa for the treatment of UTi and control of Ecoli infection
- Cran Max Sachet (Active Comparator): Cran Max is only having Vaccinium macrocarpon
  Interventions: Drug: to evaluate the safety and efficacy of Ansa for the treatment of UTi and control of Ecoli infection

INTERVENTIONS:
Drug: to evaluate the safety and efficacy of Ansa for the treatment of UTi and control of Ecoli infection — to evaluate the safety and efficacy of Cranmax for the treatment of UTi and control of Ecoli infection
  Other Names: Cranmax

SUMMARY:
I

This clinical trial aims to VIVO AND IN VITRO COMPARATIVE STUDY ON EFFICACY OF ANSA (experimental drug) & CRAN MAX (control drug) SACHET IN UNCOMPLICATED UTI in females. The main question[s] it aims to answer are:

• Hypothesis I ANSA is an effective therapy for uncomplicated UTI treatment and inhibits or kills E.coli and other organisms in vitro and in vivo Null Hypothesis ANSA is not an effective therapy for uncomplicated UTI treatment and couldn't inhibit or kill E.coli and other organisms in vitro and in vivo Hypothesis II Cran Max is an effective therapy for uncomplicated UTIs and inhibits or kills E.coli and other organisms in vitro and in vivo Null Hypothesis Cran Max is not an effective therapy for uncomplicated UTI treatment and couldn't inhibit or kill E.coli and other organisms in vitro and in vivo

DETAILED DESCRIPTION:
In this study, the emphasis is to evaluate the in vivo & in vitro efficacy of Ansa sachet having three APIs (Vaccinium macrocarpon, Saraca indica, Cimicifuga racemosa) in comparison with Cran max sachet in female patients having uncomplicated UTI. It is a single-blinded, randomized controlled trial. UTI (urinary tract infection) is mainly caused by E.coli and other associated organisms about 80% in females of fertile age and it occurs with less percentage in males. Uncommon recurrent UTIs is more prevalent in females than males. Post-menopausal women have higher rates of UTIs because of pelvic prolapse, lack of estrogen, loss of lactobacilli in the vaginal flora, increased peri-urethral colonization by Escherichia coli (E. coli), and a higher incidence of medical illnesses such as diabetes mellitus (DM).The microorganism that causes UTIs is similar, in most cases, to the sporadic infection. Most uro-pathogens from the rectal flora ascend to the bladder after colonizing in the peri urethral area and urethra. Keeping in mind that Helix Pharma designed ANSA in such a combination that it not only helps in the prevention of UTIs but also decreased recurrent UTIs as other APIs in ANSA have the capacity to normalize hormonal levels in females which is the basic cause of peri-menopausal and menopausal woman. The objective is to do a comparison of whether the Ansa sachet (experimental drug) or cran max sachet (control group) is a clinically good choice.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients of age 15 to 70 years
2. Patient suffering from complain of burning micturition and will be diagnosed as a case of uncomplicated UTI by Urine D/R
3. Female patients from Karachi related to any discipline
4. All socioeconomic classes included in the study

Exclusion Criteria:

* 1. Males are not included in this study 2. Pregnant females 3. Patient having surgical history related to renal disorder are excluded 4. Patients with co-morbidities like diabetes, uncontrolled hypertension and liver disorder are excluded 5. Patient having any drug reaction from any of the study drug is excluded 6. Patient suffering from serious illness like encephalitis, coma, meningitis or head injury are excluded

Ages: 15 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — females
Enrollment: 100 (Estimated)
Dates: Start 2021-08-12 (Actual); Primary Completion 2024-08-12 (Estimated); Study Completion 2024-08-12 (Estimated)

PRIMARY OUTCOMES:
Urine D/R | I week
  To check the urinary infection

SECONDARY OUTCOMES:
Improvement in clinical symptoms | I week
  Improvement in clinical symptoms such as burnining micturation

CONTACTS AND LOCATIONS:
Overall Officials: Misbah Ahmed, BEMS, Principal Investigator — Jinnah University
Locations (2):
- Pakistan (2):
  - Misbah Ahmed, Karachi, Sindg
  - Pakistan, Karachi, Sindh

IPD SHARING:
Plan to Share IPD: Undecided